CLINICAL TRIAL: NCT05149157
Title: Search for Correlates of Recovery in the Patient Transcriptome (SCRIPT) (Malaria) Study
Brief Title: Trajectories and Mechanisms of Recovery From Malaria: An Observational Study
Acronym: SCRIPT
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 21SM7226
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Malaria
Keywords: Malaria; Recovery; Transcriptomics
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood RNA, serum, plasma, and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Symptomatic malaria — This observational study will be recruiting patients who have symptomatic malaria (confirmed by presence of asexual stage parasitaemia of any Plasmodium species on blood film)

SUMMARY:
This observational research study aims to answer the question: 'Which aspects of human biology play an important role in recovery from symptomatic malaria?'

In particular, the researchers aim to identify human genes for which the level of gene activity reflects the patient's overall rate of recovery. The researchers believe this approach may reveal new targets for adjunctive therapies.

The researchers aim to recruit 240 people, of all ages, who have been diagnosed with symptomatic malaria at selected hospitals in London. Blood samples, urine samples, and clinical information will be collected over the 14 days following malaria diagnosis.

ELIGIBILITY:
Inclusion Criteria:

Patients of any age with symptomatic malaria confirmed by asexual stage parasitaemia (of any Plasmodium species) on blood film.

Exclusion Criteria:

Patients with asymptomatic malaria; Patients with congenital malaria; Patients with Plasmodium gametocytaemia only; Patients with known HIV; Patients who have received antimalarial treatment for symptomatic malaria in the 28 days prior to hospital presentation; Patients who explicitly deny consent.

Min Age: 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age with symptomatic malaria confirmed by asexual stage parasitaemia (of any Plasmodium species) on blood film
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Genes for which expression (level of gene activity) correlates with a 'composite recovery score' | Each study participant will be assessed over the 14 days following malaria diagnosis
  The 'composite recovery score' will be calculated by principal component analysis of rates of recovery for individual markers of tissue, organ, or organ system dysfunction, and extraction of the value of the first principal component for each participant. Genes for which expression correlates with the 'composite recovery score' will be identified by whole blood transcriptome analysis.

SECONDARY OUTCOMES:
Genes for which expression (level of gene activity) correlates with rate of recovery for individual markers of tissue, organ, or organ system dysfunction | Each study participant will be assessed over the 14 days following malaria diagnosis
  Genes for which expression correlates with the individual markers of tissue, organ, or organ system dysfunction will be identified by whole blood transcriptome analysis.
Rate of recovery for individual markers of tissue, organ, or organ system dysfunction | Each study participant will be assessed over the 14 days following malaria diagnosis
  Rates of recovery will be calculated for individual markers of tissue, organ, or organ system dysfunction
Sequences of clinical events predictive of recovery, as determined by Bayesian inference of dynamic pathways using the HyperTraPS statistical platform | Each study participant will be assessed over the 14 days following malaria diagnosis
  Hypercubic transition path sampling (HyperTraPS) will be used to characterise patterns of recovery and identify predictors of fast vs slow recovery

CONTACTS AND LOCATIONS:
Overall Officials: Aubrey Cunnington, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No